CLINICAL TRIAL: NCT00248820
Title: Contrast-Enhanced Ultrasound Ability in the Characterization of Ovarian Masses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT02-OV
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Ovarian Tumor
Keywords: Contrast-enhanced Ultrasound; Ultrasound Contrast agent, microbubbles; Ovarian tumor; vascularization
MeSH Terms: conditions — Ovarian Neoplasms; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Contrast-enhanced ultrasound — Contrast enhanced ultrasound using Sonovue / 2.4 ml per injection - one or two injections (maximum of 9.6 ml).

SUMMARY:
This study intends to assess the ability of contrast-enhanced ultrasound in the detection of benign and malignant ovarian masses compared to unenhanced ultrasound.

By using an intravascular contrast agent, this noninvasive and feasible imaging technique will allow the investigators to define specific microcirculation patterns in 100 women with ovarian lesions.

The intravascular contrast agent properties will be compared between benign and malignant adnexal masses.

The final purpose of this ultrasonography is to allow the early detection of tumors and to improve the characterization between benign and malignant lesions.

DETAILED DESCRIPTION:
SonoVue (Sulphur hexafluoride microbubbles) is a microbubbles preparation that is stable, resistant to pressure and specifically designed to be used as a contrast agent for ultrasound imaging.

Study design : one contrast-enhanced ultrasonography is proposed before any surgery to patients with ovarian mass.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient with adnexal mass detected by ultrasound
* Any programmed surgery

Exclusion Criteria:

* Any contraindication to surgery
* Injection of another contrast agent within 24 hours before the study examination
* Pregnancy, breastfeeding
* Patient known to have a coronary syndrome
* Unstable angina and myocardial infarction
* Acute cardiac failure, Class III/IV cardiac failure
* Severe rhythm disorders
* Acute endocarditis
* Prosthetic valves
* Patient previously having received an investigational drug within 30 days prior to admission into this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-09; Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
From contrast-enhanced ultrasound: Enhancement parameters derived from time-intensity curves: time-to-peak, enhancement ratio, washout-time | inclusion period

SECONDARY OUTCOMES:
Histology assessments: microvessel density assessments and histological diagnosis | inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: Henri Marret, PR, Principal Investigator — Service de Gynécologie Obstétrique - Centre Olympe de Gouges CHRU Tours; François Tranquart, PR, Study Director — Centre d'Innovation Technologique - CHRU Tours
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Background] Tailor A, Jurkovic D, Bourne TH, Collins WP, Campbell S. Sonographic prediction of malignancy in adnexal masses using multivariate logistic regression analysis. Ultrasound Obstet Gynecol. 1997 Jul;10(1):41-7. doi: 10.1046/j.1469-0705.1997.10010041.x. PMID 9263422
- [Background] MacSweeney JE, Cosgrove DO, Arenson J. Colour Doppler energy (power) mode ultrasound. Clin Radiol. 1996 Jun;51(6):387-90. doi: 10.1016/s0009-9260(96)80155-3. No abstract available. PMID 8654001
- [Background] Timmerman D, Bourne TH, Tailor A, Collins WP, Verrelst H, Vandenberghe K, Vergote I. A comparison of methods for preoperative discrimination between malignant and benign adnexal masses: the development of a new logistic regression model. Am J Obstet Gynecol. 1999 Jul;181(1):57-65. doi: 10.1016/s0002-9378(99)70436-9. PMID 10411796
- [Background] Kinkel K, Hricak H, Lu Y, Tsuda K, Filly RA. US characterization of ovarian masses: a meta-analysis. Radiology. 2000 Dec;217(3):803-11. doi: 10.1148/radiology.217.3.r00dc20803. PMID 11110947
- [Background] Suren A, Osmers R, Kulenkampff D, Kuhn W. Visualization of blood flow in small ovarian tumor vessels by transvaginal color Doppler sonography after echo enhancement with injection of Levovist. Gynecol Obstet Invest. 1994;38(3):210-2. doi: 10.1159/000292481. PMID 8001878
- [Background] Orden MR, Gudmundsson S, Kirkinen P. Contrast-enhanced sonography in the examination of benign and malignant adnexal masses. J Ultrasound Med. 2000 Nov;19(11):783-8. doi: 10.7863/jum.2000.19.11.783. PMID 11065267
- [Background] Morel DR, Schwieger I, Hohn L, Terrettaz J, Llull JB, Cornioley YA, Schneider M. Human pharmacokinetics and safety evaluation of SonoVue, a new contrast agent for ultrasound imaging. Invest Radiol. 2000 Jan;35(1):80-5. doi: 10.1097/00004424-200001000-00009. PMID 10639039